CLINICAL TRIAL: NCT06519799
Title: Integrated Genetic and Functional Analysis of the Influence of Menstrual Hygiene Products on Female Health
Acronym: Luna
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University Hospital, Antwerp (Other)
Collaborators: Universiteit Antwerpen (Other); Research Foundation Flanders (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: EDGE003611
Record Dates: First submitted 2024-05-13; First posted 2024-07-25 (Actual); Last update posted 2024-07-25 (Actual); Status verified 2024-01

CONDITIONS: Vaginal Disease; Menstrual Discomfort
Keywords: menstrual health; intimate health
MeSH Terms: conditions — Vaginal Diseases | interventions — Menstrual Hygiene Products

STUDY DESIGN:
Intervention Model Description: Each participant will wear all 5 menstrual products in a randomized order.
Masking Description: As the intervention is the use of a menstrual product, no masking is possible.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Combination pill (Experimental): This arm ( n = 50) is selected based on their contraception use, under the combination pill your menstruation and composition of menstrual blood is altered. In this arm all participants will wear all 5 menstrual products, 1 product per menstruation. The order of products will be randomized over this arm.
  Interventions: Other: Menstrual hygiene products
- No-hormonal contracteption (Experimental): This arm (n = 50) is selected based on the use of no hormonal contraception, to investigate a natural menstrual cycle. In this arm all participants will wear all 5 menstrual products, 1 product per menstruation. The order of products will be randomized over this arm.
  Interventions: Other: Menstrual hygiene products

INTERVENTIONS:
Other: Menstrual hygiene products — The influence on the intimate health of each product will be evaluated. As you can't not use a menstrual product during menstruation, no control group is included
  Other Names: Menstrual cup; tampon; Menstrual pad; Menstrual underwear with cotton crotch; Menstrual underwear with non-cotton crotch

SUMMARY:
Women's reproductive health has attracted increasing attention in recent years, including in the field of microbiology. Vaginal infections, such as vulvovaginal candidiasis, bacterial vaginosis and aerobic vaginitis, are common and a huge burden on our society. The vaginal microbiome is important in the prevention of these infections, in fertility and for healthy pregnancies. The composition, and therefore the 'health' of the vaginal microbiome, is influenced by many internal and external factors, including intimate health. However, it is not yet known how intimate health, and specifically the use of menstrual hygiene products, affects the microbiome and women's intimate comfort and health. In this study, the researchers aim to understand the influence of 5 menstrual hygiene products (tampon, menstrual cup, menstrual pad and 2 types of menstrual underwear) on women's intimate health (n = 100). First, this will be evaluated at the microbiome level, focusing on the female intimate microbiome, consisting of the skin in the groin, vulvar and vaginal microbiome. These sites are all closely linked and are affected in vaginal infections or by contact with menstrual hygiene products. Second, in addition to the direct impact on the microbiome, the impact on the participant's immune system will be evaluated, as some well-known menstrual hygiene products can cause irritation and inflammation. As a third goal, participants will assess the comfort and usability of each menstrual hygiene product and provide data on their lifestyle and other factors that may influence our results. The main goal is to investigate and define the impact of menstrual hygiene products on women's intimate health so that women can make an informed choice. In a first phase participants (n = 1500) will fill in a survey containing questions on general health, lifestyle and menstrual health. Based on these responses a selection of 100 participants will be made by the researchers to participate in the intervention trial.

ELIGIBILITY:
Inclusion Criteria:

* female
* contraception: combination pill with stop week or no hormonal contraception
* premenopausal
* Dutch-speaking living in Belgium
* regular menstrual cycle (if no hormonal contraception)

Exclusion Criteria:

* Pregnancy

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — people who menstruate
Enrollment: 100 (Estimated)
Dates: Start 2024-08-01 (Estimated); Primary Completion 2025-02-01 (Estimated); Study Completion 2025-10-31 (Estimated)

PRIMARY OUTCOMES:
Beta diversity of the vaginal microbiome | Each month for 3 samplepoints until study completion, an average of 6 months
  This measure describes the taxonomic diversity between samples, a higher diversity is associated with a less healthy vaginal microbiome. Beta diversity within a participant over all products will be calculated as a stability measure. This will be defined for each participant comparing the baseline samples (right before menstruation) to the sample during and after menstruation. Comparison will be made between different menstrual hygiene products.

SECONDARY OUTCOMES:
relative abundance of eigentaxa | Each month for 3 samplepoints until study completion, an average of 6 months
  The relative abundance of some eigentaxa such as Lactobacillus crispatus will be looked at, as this is known to be associated with some menstrual products. The relative abundance at each samplepoint will be evaluated at the end of the study, comparison will be made between the different menstrual hygiene products.
comfort and ease of use | Periodically, after menstruation once a month.
  the participants will answer evaluate the comfort and ease of use of each product, during the survey at the timepoint after each menstruation for each product.
alfa diversity of the vaginal microbiome | Each month for 3 samplepoints until study completion, an average of 6 months
  this measure describes the taxonomic diversity within a sample. The alfa diversity within a participant over all products will be calculated as a measure of stability. This will be defined for each participant comparing the baseline samples (right before menstruation) to the sample during and after menstruation. Comparison will be made between different menstrual hygiene products.
both alfa and beta diversity of the vulvar and groin skin microbiome | Each month for 3 samplepoints until study completion, an average of 6 months
  these measures describe the taxonomic diversity. Comparison will be made between different menstrual hygiene products.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Antwerp, Antwerp, Belgium

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (2):
  • Study Protocol (2023-12-21): https://cdn.clinicaltrials.gov/large-docs/99/NCT06519799/Prot_000.pdf
  • Informed Consent Form (2024-05-13): https://cdn.clinicaltrials.gov/large-docs/99/NCT06519799/ICF_001.pdf